CLINICAL TRIAL: NCT03530917
Title: A Randomized, Sponsor-Open, Investigator-Blinded, Subject-Blinded, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7020531 and Metabolites Following Oral Administration to Chinese Healthy Volunteers.
Brief Title: A Study to Assess the Safety and Tolerability of Single and Multiple Ascending Doses of Oral RO7020531 in Chinese Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: YP39553
Record Dates: First submitted 2018-05-09; First posted 2018-05-21 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Healthy Participants
MeSH Terms: interventions — RO7020531

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Single Ascending Dose (SAD): Placebo (Experimental): In SAD Cohorts 1-4, there will be eight participants in total receiving placebo, two in each cohort.
  Interventions: Drug: Placebo
- SAD: Cohort 1 (Experimental): Eight participants will be administered 40mg RO7020531 orally on Day 1.
  Interventions: Drug: RO7020531
- SAD: Cohort 2 (Experimental): Eight participants will be administered 100mg RO7020531 orally on Day 1.
  Interventions: Drug: RO7020531
- SAD: Cohort 3 (Experimental): Eight participants will be administered 140mg RO7020531 orally on Day 1.
  Interventions: Drug: RO7020531
- SAD: Cohort 4 (Experimental): Eight participants will be administered 170mg RO7020531 orally on Day 1.
  Interventions: Drug: RO7020531
- Multiple Ascending Dose (MAD): Placebo (Experimental): In MAD Cohorts 1-3, there will be six participants in total receiving placebo, two in each cohort.
  Interventions: Drug: Placebo
- MAD: Cohort 1 (Experimental): Eight participants will be administered 100mg RO7020531 orally on Day 1 and every other day (QOD) for 14 days.
  Interventions: Drug: RO7020531
- MAD: Cohorts 2 and 3 (Experimental): Sixteen participants will be administered 150mg RO7020531 orally on Day 1 and every other day (QOD) for 14 days.
  Interventions: Drug: RO7020531

INTERVENTIONS:
Drug: RO7020531 — 4 SAD Cohorts with individual dosages of 40, 100, 140 and 170 mg hard capsules and 3 MAD Cohorts with dosages of 100 and 150mg hard capsules, will be administered orally as per the dosing schedules described above.
  Arms: MAD: Cohort 1; MAD: Cohorts 2 and 3; SAD: Cohort 1; SAD: Cohort 2; SAD: Cohort 3; SAD: Cohort 4
Drug: Placebo — Placebo hard capsules will be administered orally as per the dosing schedules described above.
  Arms: Multiple Ascending Dose (MAD): Placebo; Single Ascending Dose (SAD): Placebo

SUMMARY:
To evaluate the safety and tolerability of single and multiple ascending doses of oral RO7020531 in Chinese healthy participants.

ELIGIBILITY:
Inclusion Criteria

* Chinese healthy male and female participants. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, and urinalysis.
* A Body Mass Index (BMI) of 19 to less than 28 kg/m2 and a body weight of at least 45 kg.
* Negative anti-nuclear antibody (ANA) test; or positive with dilutions not greater than 1:40 and with no associated history or symptoms of potential connective tissue disease or other immune-mediated diseases.
* Women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods.
* Men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and refrain from donating sperm.
* Negative pregnancy test on Day -1 for female participants.
* Non-smokers, or use of < 10 cigarettes (or equivalent nicotine-containing product) per day.

Exclusion Criteria

* Pregnant (positive pregnancy test) or lactating women, and male partners of women who are pregnant or lactating.
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis, multiple sclerosis, or any other autoimmune disease).
* History or symptoms of any clinically significant disease including (but not limited to), neurological, cardiovascular, endocrine, respiratory, hepatic, ocular, or renal disorder (as per Investigator's judgment).
* Personal or family history of congenital long QT syndrome or sudden cardiac death.
* Evidence of an active or suspected cancer or a history of malignancy, where in the Investigator's opinion, there is a risk of recurrence.
* History of having received or currently receiving any systemic anti-neoplastic (including radiation) or immune-modulatory treatment (including systemic oral or inhaled corticosteroids, IFN or PEG-IFN) within 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study. Eye drop-containing and infrequent inhaled corticosteroids are permissible up to 4 weeks prior to the first dose of study drug.
* History of clinically significant thyroid disease; also, subjects with clinically significant elevated thyroid-stimulating hormone (TSH) concentrations at Screening.
* Any confirmed clinically significant allergic reactions (anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable).
* Abnormal renal function.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values at Screening above ULN and judged clinically significant by the Investigator.
* Positive results for anti-mitochondrial antibody (AMA), anti-smooth muscle antibody (ASMA) or thyroid peroxidase antibody.
* Positive hepatitis A IgM antibody (HAV Ab IgM), hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or positive for human immunodeficiency virus (HIV) at Screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 Center in China.
Pre-assignment Details: A total of 70 Healthy Male and Female Chinese Participants were enrolled.
Period: Overall Study
Arm/Group | Single Ascending Dose (SAD): Placebo | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | Multiple Ascending Dose (MAD): Placebo | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Started | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
Completed | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Ascending Dose (SAD): Placebo | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | Multiple Ascending Dose (MAD): Placebo | MAD: Cohort 1 | MAD: Cohorts 2 and 3 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.25 (6.65) | 25.25 (7.67) | 24.13 (8.58) | 23.00 (3.66) | 26.75 (9.44) | 22.50 (3.02) | 25.75 (8.24) | 23.19 (3.37) | 24.50 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 1 | 4 | 2 | 2 | 4 | 3 | 25
  Male | 4 | 3 | 7 | 4 | 6 | 4 | 4 | 13 | 45
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, any deterioration in a laboratory value or other clinical test or adverse events that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment.
Time Frame: Screening up until 28 days after the last dose of study drug (up to 1 year).
Population: The Safety Population was defined as all Healthy Volunteers who have received at least one dose of the study medication, whether prematurely withdrawn from the study or not.
Measure: Number; unit: Percentage of Participants
Arm/Group | Single Ascending Dose (SAD): Placebo | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | Multiple Ascending Dose (MAD): Placebo | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
Percentage of Participants | 37.5 | 37.5 | 25.0 | 50.0 | 100 | 100 | 100 | 93.8

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for RO7020531, Main Active Metabolite (RO7011785) and Prodrug Metabolites (RO7018822 and RO7033805)
Description: Non-compartmental analysis using WinNonlin software was used to calculate PK parameters where appropriate. Summary descriptive statistics (Arithmetic Mean and Standard Deviation) for Cmax will be presented by treatment arm. Where appropriate, data maybe pooled and analyzed. Please note that this Outcome Measure was not measured for the Placebo Cohorts and SAD Cohorts (1-4) (on Day 13).
Time Frame: SAD: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48 hours (h) Post-dose Days 1, 2; MAD: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24h Post-dose Days 1, 2 and Days 13, 14; Pre-dose, 2, 6, 24hr Post-dose Days 3, 5, 7, 9 and 11.
Population: The PK analysis population included all healthy volunteers randomised and adherent to the protocol. Participants were excluded if they significantly violated the inclusion/exclusion criteria, deviated significantly from the protocol or if data were unavailable or incomplete. Data presented is only for participants included in the actual analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 16
ng/ml
  Day 1 (RO7020531): number analyzed (Participants) | 8 | 8 | 8 | 8 | 0 | 1
  Day 1 (RO7020531) | NA (NA) — Values were below the lower limit of quantification. | NA (NA) — Values were below the lower limit of quantification. | 0.14 (0.39) | NA (NA) — Values were below the lower limit of quantification. |  | 1.08 (NA) — Values were below the lower limit of quantification.
  Day 13 (RO7020531): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Day 13 (RO7020531) |  |  |  |  |  | 1.56 (NA) — Values were below the lower limit of quantification.
  Day 1 (RO7011785) | 640 (227) | 1380 (461) | 1940 (516) | 2180 (841) | 1290 (414) | 1900 (501)
  Day 13 (RO7011785): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
  Day 13 (RO7011785) |  |  |  |  | 1110 (480) | 1530 (382)
  Day 1 (RO7018822) | 78.6 (32.9) | 125 (56.7) | 200 (70.4) | 247 (112) | 249 (217) | 231 (98.5)
  Day 13 (RO7018822): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
  Day 13 (RO7018822) |  |  |  |  | 116 (55.2) | 155 (50.6)
  Day 1 (RO7033805): number analyzed (Participants) | 8 | 8 | 8 | 8 | 0 | 0
  Day 1 (RO7033805) | NA (NA) — Values were below the lower limit of quantification. | NA (NA) — Values were below the lower limit of quantification. | 0.14 (0.39) | NA (NA) — Values were below the lower limit of quantification. |  |
  Day 13 (RO7033805): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Day 13 (RO7033805) |  |  |  |  |  | 1.08 (NA) — Values were below the lower limit of quantification.

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve up to the Last Measurable Concentration (AUClast) for RO7020531, Main Active Metabolite (RO7011785) and Prodrug Metabolites (RO7018822 and RO7033805)
Description: Non-compartmental analysis using WinNonlin software was used to calculate PK parameters where appropriate. Summary descriptive statistics (Arithmetic Mean and Standard Deviation) for AUClast will be presented by treatment arm. Where appropriate, data maybe pooled and analyzed. Please note that this Outcome Measure was not measured for the Placebo Cohorts and SAD Cohorts (1-4) (on Day 13).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 16
hr*ng/ml
  Day 1 (RO7020531): number analyzed (Participants) | 8 | 8 | 8 | 8 | 0 | 1
  Day 1 (RO7020531) | 0.00 (0.00) | 0.00 (0.00) | 0.02 (0.05) | 0.00 (0.00) |  | 0.14 (NA) — Values were below the lower limit of quantification.
  Day 13 (RO7020531): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Day 13 (RO7020531) |  |  |  |  |  | 0.92 (NA) — Values were below the lower limit of quantification.
  Day 1 (RO7011785) | 707 (155) | 1660 (229) | 2500 (550) | 2700 (467) | 1870 (333) | 2650 (389)
  Day 13 (RO7011785): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
  Day 13 (RO7011785) |  |  |  |  | 1650 (313) | 2550 (521)
  Day 1 (RO7018822) | 57.9 (22.8) | 109 (29.7) | 199 (78.9) | 250 (125) | 235 (125) | 211 (58.5)
  Day 13 (RO7018822): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
  Day 13 (RO7018822) |  |  |  |  | 169 (98.8) | 184 (51.0)
  Day 1 (RO7033805): number analyzed (Participants) | 8 | 8 | 8 | 8 | 0 | 0
  Day 1 (RO7033805) | 0.00 (0.00) | 0.00 (0.00) | 0.02 (0.05) | 0.00 (0.00) |  |
  Day 13 (RO7033805): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Day 13 (RO7033805) |  |  |  |  |  | 0.14 (NA) — Values were below the lower limit of quantification.

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUCinf) for RO7020531, Main Active Metabolite (RO7011785) and Prodrug Metabolites (RO7018822 and RO7033805)
Description: Non-compartmental analysis using WinNonlin software was used to calculate PK parameters where appropriate. Summary descriptive statistics (Arithmetic Mean and Standard Deviation) for AUCinf will be presented by treatment arm. Where appropriate, data maybe pooled and analyzed. Please note that this Outcome Measure was not measured for the Placebo Cohorts and SAD Cohorts (1-4) (on Day 13). Due to insufficient plasma concentration data for RO7020531 and RO7033805, AUCinf for these 2 compounds could not be estimated.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 16
hr*ng/ml
  Day 1 (RO7020531): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Day 13 (RO7020531): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 (RO7011785) | 714 (154) | 1670 (229) | 2510 (549) | 2720 (467) | 1880 (333) | 2660 (389)
  Day 13 (RO7011785): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
  Day 13 (RO7011785) |  |  |  |  | 1660 (311) | 2510 (523)
  Day 1 (RO7018822): number analyzed (Participants) | 8 | 8 | 8 | 7 | 7 | 16
  Day 1 (RO7018822) | 58.5 (22.8) | 111 (29.6) | 204 (80.6) | 245 (133) | 241 (135) | 214 (58.7)
  Day 13 (RO7018822): number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 8
  Day 13 (RO7018822) |  |  |  |  | 177 (115) | 189 (52.4)
  Day 1 (RO7033805): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Day 13 (RO7033805): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for RO7020531, Main Active Metabolite (RO7011785) and Prodrug Metabolites (RO7018822 and RO7033805)
Description: Non-compartmental analysis using WinNonlin software was used to calculate PK parameters where appropriate. Summary descriptive statistics (Median and Full Range) for Tmax will be presented by treatment arm. Where appropriate, data maybe pooled and analyzed. Please note that this Outcome Measure was not measured for the Placebo Cohorts and SAD Cohorts (1-4) (on Day 13).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 16
hr
  Day 1 (RO7020531): number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  Day 1 (RO7020531) |  |  | 0.50 [0.5 to 0.5] |  |  | 0.25 [0.25 to 0.25]
  Day 13 (RO7020531): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Day 13 (RO7020531) |  |  |  |  |  | 0.50 [0.5 to 0.5]
  Day 1 (RO7011785) | 0.50 [0.50 to 1.00] | 0.75 [0.50 to 1.50] | 0.50 [0.50 to 1.50] | 0.50 [0.50 to 1.50] | 1.50 [0.50 to 2.00] | 0.52 [0.50 to 1.50]
  Day 13 (RO7011785): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
  Day 13 (RO7011785) |  |  |  |  | 1.00 [0.53 to 3.00] | 1.00 [0.50 to 1.50]
  Day 1 (RO7018822) | 0.50 [0.50 to 1.00] | 0.50 [0.25 to 1.50] | 0.50 [0.25 to 1.50] | 0.50 [0.50 to 2.00] | 0.50 [0.25 to 2.00] | 0.50 [0.25 to 1.50]
  Day 13 (RO7018822): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
  Day 13 (RO7018822) |  |  |  |  | 1.00 [0.25 to 3.00] | 0.50 [0.50 to 1.50]
  Day 1 (RO7033805): number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  Day 1 (RO7033805) |  |  | 0.50 [0.5 to 0.5] |  |  |
  Day 13 (RO7033805): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Day 13 (RO7033805) |  |  |  |  |  | 0.50 [0.5 to 0.5]

6. Secondary Outcome: Half-Life (t1/2) for RO7020531, Main Active Metabolite (RO7011785) and Prodrug Metabolites (RO7018822 and RO7033805)
Description: Non-compartmental analysis using WinNonlin software was used to calculate PK parameters where appropriate. Summary descriptive statistics (Arithmetic Mean and Standard Deviation) for t1/2 will be presented by treatment arm. Where appropriate, data maybe pooled and analyzed. Please note that this Outcome Measure was not measured for the Placebo Cohorts and SAD Cohorts (1-4) (on Day 13). Due to insufficient plasma concentration data for RO7020531 and RO7033805, t1/2 for these 2 compounds could not be estimated.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 16
hr
  Day 1 (RO7020531): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Day 13 (RO7020531): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 (RO7011785) | 2.92 (0.787) | 3.38 (0.499) | 3.96 (0.761) | 4.24 (0.667) | 3.38 (0.976) | 4.39 (0.918)
  Day 13 (RO7011785): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8
  Day 13 (RO7011785) |  |  |  |  | 3.52 (0.813) | 3.85 (0.807)
  Day 1 (RO7018822): number analyzed (Participants) | 8 | 8 | 8 | 7 | 7 | 16
  Day 1 (RO7018822) | 0.519 (0.124) | 0.606 (0.0932) | 0.642 (0.160) | 0.612 (0.172) | 0.605 (0.0920) | 0.611 (0.0935)
  Day 13 (RO7018822): number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 8
  Day 13 (RO7018822) |  |  |  |  | 0.753 (0.189) | 0.706 (0.315)
  Day 1 (RO7033805): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Day 13 (RO7033805): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Total Amount Excreted as RO7020531, RO7011785, RO7018822 and RO7033805
Description: Non-compartmental analysis using WinNonlin software was used to calculate PK parameters where appropriate. Summary descriptive statistics (Arithmetic Mean and Standard Deviation) for Total Amount Excreted, will be presented by treatment arm. Where appropriate, data maybe pooled and analyzed. Please note that this Outcome Measure was not measured for the Placebo Cohorts and MAD Cohorts (1-4).
Time Frame: SAD: Pre-dose, 0-4, 4-8, 8-12, 12-24h Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4
Number analyzed (Participants) | 8 | 8 | 8 | 8
mg
  RO7020531: number analyzed (Participants) | 8 | 8 | 2 | 0
  RO7020531 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |
  RO7011785 | 22.2 (1.96) | 58.3 (6.27) | 87.0 (10.1) | 104 (14.9)
  RO7018822 | 0.39 (0.14) | 0.74 (0.16) | 1.31 (0.40) | 1.63 (0.51)
  RO7033805: number analyzed (Participants) | 8 | 8 | 2 | 0
  RO7033805 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |

8. Secondary Outcome: Fraction Excreted as RO7020531, RO7011785, RO7018822 and RO7033805
Description: Non-compartmental analysis using WinNonlin software was used to calculate PK parameters where appropriate. Summary descriptive statistics (Arithmetic Mean and Standard Deviation) for Fraction Excreted (Molecular Weight corrected) will be presented by treatment arm. Where appropriate, data maybe pooled and analyzed. Please note that this Outcome Measure was not measured for the Placebo Cohorts and MAD Cohorts (1-4).
Time Frame: SAD: Pre-dose, 0-4, 4-8, 8-12, 12-24h Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4
Number analyzed (Participants) | 8 | 8 | 8 | 8
Percentage
  RO7020531: number analyzed (Participants) | 8 | 8 | 2 | 0
  RO7020531 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |
  RO7011785 | 59.9 (5.30) | 62.9 (6.77) | 67.1 (7.78) | 66.2 (9.47)
  RO7018822 | 1.10 (0.40) | 0.84 (0.18) | 1.06 (0.33) | 1.09 (0.34)
  RO7033805: number analyzed (Participants) | 8 | 8 | 2 | 0
  RO7033805 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |

9. Secondary Outcome: Renal Clearance of RO7020531, RO7011785, RO7018822 and RO7033805
Description: Non-compartmental analysis using WinNonlin software was used to calculate PK parameters where appropriate. Summary descriptive statistics (Arithmetic Mean and Standard Deviation) for Renal Clearance will be presented by treatment arm. Where appropriate, data maybe pooled and analyzed. Please note that this Outcome Measure was not measured for the Placebo Cohorts and MAD Cohorts (1-4). Due to insufficient urine concentration data for RO7020531 and RO7033805, Renal Clearance for these 2 compounds could not be estimated.
Time Frame: SAD: Pre-dose, 0-4, 4-8, 8-12, 12-24h Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: CLr (mL/min)
Arm/Group | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4
Number analyzed (Participants) | 8 | 8 | 8 | 8
CLr (mL/min)
  RO7020531: number analyzed (Participants) | 0 | 0 | 0 | 0
  RO7011785 | 536 (101) | 590 (78.4) | 600 (136) | 659 (157)
  RO7018822: number analyzed (Participants) | 8 | 8 | 8 | 7
  RO7018822 | 115.31 (48.54) | 116.30 (36.41) | 117.80 (42.15) | 119.99 (36.54)
  RO7033805: number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Mean Concentrations of Protein and Metabolite Markers of Humoral Response
Description: Protein and metabolite markers of humoral response include interferon (IFN)-alfa, IP-10, Tumor Necrosis Factor (TNF)-alfa, interleukin (IL)-6, IL-10, IL-12p40 and Neopterin. Summary descriptive statistics will be presented for the induction of cytokines, chemokines and neopterin and of interferon-response genes separately by treatment arm. Only mean concentrations were collected for IFN-alfa and hence why this data is only presented below.
Time Frame: SAD: Day -1, Pre-dose, 2, 6, 12, 24h Post-dose Day 1 to Day 2, 3, 5, 8; MAD: Day -1, Pre-dose 2, 6, 12, 24h Post-dose Day 1 to Day 2, Pre-dose, 2, 6, 24h Post-dose Days 3, 5, 7, 13 and 20
Population: The Pharmacodynamic (PD) analysis population was defined as all participants who were randomized, received at least one dose of study medication (RO7020531 or placebo), and have PD data available.
Measure: Geometric Mean (Standard Deviation); unit: ng/L
Arm/Group | Single Ascending Dose (SAD): Placebo | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | Multiple Ascending Dose (MAD): Placebo | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
ng/L | 0.1232 (8.5366) | 0.0433 (1.0244) | 0.0707 (2.3422) | 0.1316 (3.6720) | 0.1156 (3.6654) | 0.0455 (1.2143) | 0.1339 (4.1386) | 0.3733 (6.4327)

11. Secondary Outcome: Mean Fold Changes of Protein and Metabolite Markers of Humoral Response
Description: Protein and metabolite markers of humoral response include interferon (IFN)-alfa, IP-10, Tumor Necrosis Factor (TNF)-alfa, interleukin (IL)-6, IL-10, IL-12p40 and Neopterin. Summary descriptive statistics will be presented for the induction of cytokines, chemokines and neopterin and of interferon-response genes separately by treatment arm. Mean fold change data is presented below.
Time Frame: SAD: Day -1, Pre-dose, 2, 6, 12, 24, 48 (only Neopterin), 96h (only Neopterin), Post-dose Day 1 to Day 2, 3, 5, 8; MAD: Day -1, Pre-dose 2, 6, 12, 24h Post-dose Day 1 to Day 2, Pre-dose, 2, 6, 24h Post-dose Days 3, 5, 7, 13 and 20
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: Fold Change
Arm/Group | Single Ascending Dose (SAD): Placebo | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | Multiple Ascending Dose (MAD): Placebo | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
Fold Change
  IP-10 | 1.1108 [0.589 to 2.088] | 0.9522 [0.651 to 1.552] | 0.9987 [0.265 to 4.637] | 1.5327 [0.570 to 7.885] | 1.6229 [0.607 to 25.958] | 0.8087 [0.191 to 2.084] | 1.4014 [0.545 to 21.149] | 2.1550 [0.374 to 49.901]
  Neopterin | 1.0757 [0.741 to 1.766] | 1.0175 [0.759 to 1.287] | 1.0408 [0.621 to 1.783] | 1.1615 [0.811 to 3.000] | 1.2142 [0.824 to 3.561] | 0.9003 [0.278 to 1.750] | 1.2012 [0.754 to 3.071] | 1.6792 [0.445 to 7.797]
  Tumor Necrosis Factor (TNF)-alfa | 1.0233 [0.664 to 2.027] | 0.9286 [0.480 to 1.877] | 0.7816 [0.054 to 2.153] | 1.2098 [0.563 to 2.187] | 1.0947 [0.507 to 3.196] | 0.7482 [0.086 to 1.881] | 0.9661 [0.064 to 2.375] | 0.9909 [0.170 to 2.591]
  IL-6 | 1.0699 [0.208 to 2.719] | 0.9374 [0.223 to 2.676] | 1.0253 [0.105 to 8.919] | 1.1300 [0.483 to 2.975] | 1.0363 [0.273 to 4.513] | 0.8815 [0.059 to 8.506] | 1.0762 [0.304 to 9.522] | 1.0702 [0.081 to 10.878]
  IL-10 | 0.9410 [0.390 to 1.757] | 0.8394 [0.388 to 2.571] | 1.0561 [0.317 to 4.244] | 1.0567 [0.860 to 1.847] | 1.1666 [0.679 to 3.834] | 0.8262 [0.074 to 10.016] | 0.9641 [0.083 to 3.116] | 0.9662 [0.138 to 5.398]
  IL-12p40 | 0.9126 [0.296 to 1.504] | 0.9872 [0.749 to 2.252] | 0.9844 [0.470 to 2.971] | 0.9811 [0.863 to 1.289] | 0.9781 [0.658 to 1.536] | 1.0260 [1.000 to 1.792] | 0.9384 [0.386 to 5.008] | 1.0331 [1.000 to 2.311]

12. Secondary Outcome: Mean Fold Changes of Markers of Transcriptional Responses
Description: Markers of transcriptional responses includes ISG15, OAS-1, MX1 and Toll-Like Receptor (TLR)7. Summary descriptive statistics will be presented for these markers separately by treatment arm.
Time Frame: SAD: Day -1, Pre-dose, 2, 6, 12, 24h Post-dose Day 1 to Day 2 and Day 8; MAD: Day -1, Pre-dose 2, 6, 12, 24h Post-dose Day 1 to Day 2, Pre-dose, 2, 6, 24h Post-dose Days 3, 5, 7, 13 and 20
Population: The PD analysis population was defined as all participants who were randomized, received at least one dose of study medication (RO7020531 or placebo), and have PD data available.
Measure: Geometric Mean (Full Range); unit: Fold Change
Arm/Group | Single Ascending Dose (SAD): Placebo | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | Multiple Ascending Dose (MAD): Placebo | MAD: Cohort 1 | MAD: Cohorts 2 and 3
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 6 | 8 | 16
Fold Change
  ISG15 mRNA | 1.0538 [0.097 to 2.471] | 1.0907 [0.381 to 2.255] | 1.9190 [0.404 to 16.973] | 4.0828 [0.272 to 119.203] | 4.3223 [0.522 to 49.787] | 0.6938 [0.043 to 18.505] | 2.0720 [0.284 to 66.544] | 4.2679 [0.108 to 285.243]
  OAS-1 mRNA | 1.0739 [0.240 to 1.948] | 1.1256 [0.689 to 1.723] | 1.6148 [0.445 to 8.118] | 2.9338 [0.273 to 18.984] | 3.0716 [0.908 to 21.051] | 0.6315 [0.065 to 3.918] | 1.9447 [0.400 to 30.905] | 3.1327 [0.242 to 84.463]
  MX1 mRNA | 1.0562 [0.158 to 2.544] | 1.1742 [0.506 to 1.848] | 2.1984 [0.536 to 12.948] | 3.8705 [0.299 to 46.893] | 4.3748 [0.784 to 46.515] | 0.7414 [0.066 to 6.957] | 1.8317 [0.312 to 30.016] | 3.0186 [0.183 to 106.211]
  TLR7 mRNA | 1.0883 [0.258 to 2.595] | 1.1638 [0.587 to 2.301] | 0.9921 [0.471 to 3.214] | 2.0835 [0.602 to 11.521] | 1.3872 [0.299 to 4.584] | 0.8483 [0.275 to 1.708] | 1.4923 [0.442 to 6.572] | 1.5454 [0.243 to 17.387]

ADVERSE EVENTS:
Time Frame: Screening up until 28 days after the last dose of study drug (up to 1 year).
Description: The Safety Population was defined as all Healthy Volunteers who have received at least one dose of the study medication, whether prematurely withdrawn from the study or not. AEs that were entered into the database at the time of the database lock were included in the AE analysis.
Arm/Group | Single Ascending Dose (SAD): Placebo | SAD: Cohort 1 | SAD: Cohort 2 | SAD: Cohort 3 | SAD: Cohort 4 | Multiple Ascending Dose (MAD): Placebo | MAD: Cohort 1 | MAD: Cohorts 2 and 3
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/6 | 0/8 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 1/8 | 0/6 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 3/8 | 3/8 | 2/8 | 4/8 | 7/8 | 6/6 | 8/8 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Ascending Dose (SAD): Placebo (N=8) | SAD: Cohort 1 (N=8) | SAD: Cohort 2 (N=8) | SAD: Cohort 3 (N=8) | SAD: Cohort 4 (N=8) | Multiple Ascending Dose (MAD): Placebo (N=6) | MAD: Cohort 1 (N=8) | MAD: Cohorts 2 and 3 (N=16)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Ascending Dose (SAD): Placebo (N=8) | SAD: Cohort 1 (N=8) | SAD: Cohort 2 (N=8) | SAD: Cohort 3 (N=8) | SAD: Cohort 4 (N=8) | Multiple Ascending Dose (MAD): Placebo (N=6) | MAD: Cohort 1 (N=8) | MAD: Cohorts 2 and 3 (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Catheter site bruise (General disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Catheter site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03530917/Prot_SAP_000.pdf